CLINICAL TRIAL: NCT02228356
Title: Non-interventional Observational Study of Stereotactic Body Radiotherapy (SBRT) for Oligometastatic Cancer
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Universitair Ziekenhuis Brussel (Other)
Responsible Party: Principal Investigator, Benedikt Engels, MD, PhD, Radiation Oncologist, Universitair Ziekenhuis Brussel
Other Study IDs: BUN143201215117; BUN143201215117 (Registry Identifier: UZ Brussel Ethics Committee)
Record Dates: First submitted 2014-08-22; First posted 2014-08-29 (Estimated); Last update posted 2016-05-11 (Estimated); Status verified 2016-05

CONDITIONS: Neoplasm Metastasis
Keywords: Neoplasm Metastasis; oligometastatic cancer; Stereotactic Body Radiation Therapy; SBRT; Real-time Tumor Tracking (RTTT); ITV; Internal Target Volume; Respiratory Motion Management; Image-guided Radiotherapy; IGRT
MeSH Terms: conditions — Neoplasm Metastasis | interventions — Radiosurgery; Radiotherapy, Intensity-Modulated

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

INTERVENTIONS:
Radiation: Stereotactic Body Radiation Therapy — Stereotactic Body Radiation Therapy with either Dynamic Tumor Tracking/Internal Target Volume approach on the Vero machine, and/or Internal Target Volume approach on the Tomotherapy machine.
  Other Names: Vero; Tomotherapy

SUMMARY:
The investigators recently published 2 phase II trials on the use of helical tomotherapy for oligometastatic colorectal cancer [1,2]. Despite a dose increase from 40 to 50 Gy, delivered in 2 weeks time, the one-year local control was 54% only [1,2]. The high local failure rate is probably the result of geographical misses due to tumor motion and a biologically effective dose (BED) of < 100 Gy. The current study will investigate whether the one-year local control rate can be improved to 70%, using respiration correlated CT to individualize the margin needed to account for tumor motion, to avoid geographical miss, together with a Monte Carlo or collapsed cone dose calculation algorithm delivering 50 Gy to the 80% isodose, allowing higher doses in the tumor core. As the concept of an internal target volume (ITV) may result in large margins for patients displaying metastases in high mobile organs, such as liver and lung, which may lead to exposure of a relatively high dose to a large volume of normal tissue, dynamic tumor tracking by the VERO SBRT system will be applied in those patients.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with metastatic cancer from any primary origin and no more than 5 metastases on CT--scan
2. Primary tumor treated with curative intention (surgery, radiotherapy, chemoradiotherapy)
3. Functional liver volume > 1000cc in case of liver metastases and a lung diffusion capacity for carbon monoxide (DLCO) of > 30% if lung mets
4. No Child B or C liver cirrhosis
5. No systemic treatment within 1 month before initiation of radiotherapy
6. No contra-indications for radiation of all metastatic disease (= no violation of constraints of organs at risk (OAR))
7. No metastases from another carcinoma
8. Eastern Cooperative Oncology Group (ECOG) performance status ≤ 2
9. Age > 18 years

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with metastatic cancer from any primary origin and no more than 5 metastases.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2012-06; Primary Completion 2017-06 (Estimated)

PRIMARY OUTCOMES:
One year local control | one year post radiotherapy

SECONDARY OUTCOMES:
Acute toxicity | Up to 3 months post radiotherapy
Survival | 3 to 36 months post Radiotherapy
  Overall survival
Progression Free Survival | 3 to 36 months post Radiotherapy
Late toxicity | 3 to 36 months post Radiotherapy

CONTACTS AND LOCATIONS:
Overall Officials: Benedikt Engels, MD, PhD, Principal Investigator — Dienst Radiotherapie, UZ Brussel, Vrije Universiteit Brussel; Robbe Van den Begin, MD, Principal Investigator — Dienst Radiotherapie, UZ Brussel, Vrije Universiteit Brussel; Mark De Ridder, MD, PhD, Principal Investigator — Dienst Radiotherapie, UZ Brussel, Vrije Universiteit Brussel
Locations (1):
- UZ Brussel Radiotherapie dienst, Jette, Brussels Capital, Belgium

REFERENCES:
- [Background] Engels B, Everaert H, Gevaert T, Duchateau M, Neyns B, Sermeus A, Tournel K, Verellen D, Storme G, De Ridder M. Phase II study of helical tomotherapy for oligometastatic colorectal cancer. Ann Oncol. 2011 Feb;22(2):362-8. doi: 10.1093/annonc/mdq385. Epub 2010 Aug 4. PMID 20685718
- [Background] Engels B, Gevaert T, Everaert H, De Coninck P, Sermeus A, Christian N, Storme G, Verellen D, De Ridder M. Phase II study of helical tomotherapy in the multidisciplinary treatment of oligometastatic colorectal cancer. Radiat Oncol. 2012 Mar 16;7:34. doi: 10.1186/1748-717X-7-34. PMID 22423615